CLINICAL TRIAL: NCT05208151
Title: The Perceived Effect of Communication Skills Education Integrated With Creative Drama on Physiotherapy and Rehabilitation Students' Empathy and Communication Skills to Develop With the Patient: A Randomized Controlled Study
Brief Title: Creative Drama in Physiotherapy and Rehabilitation Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc Prof. Nuray Alaca, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ATADEK-2021/22/06
Record Dates: First submitted 2021-12-28; First posted 2022-01-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Educational Problems
Keywords: Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative Drama Group (Active Comparator)
  Interventions: Other: Creative Drama Education
- Control Group (No Intervention)

INTERVENTIONS:
Other: Creative Drama Education — Effective Communication with Creative Drama in Health Course will be given to students for 2 hours a week for 14 weeks.
  Arms: Creative Drama Group

SUMMARY:
Candidates who will provide the health services of the future should be ready to provide the safe and best health care services. In order to achieve this, it is recommended to use new training programs and methods that will provide similar situations to the working environment in the training of health workers. There are very few studies on the empathy and communication perceptions that creative drama education will create with the patient on physiotherapy and rehabilitation department students. Therefore, this study, the investigators aimed to investigate the perceived effect of communication skills training integrated with creative drama on physiotherapy and rehabilitation students' empathy and communication skills that will develop with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to take FZT 233 Effective Communication with Creative Drama in Health course in any of the fall or spring semesters.

Exclusion Criteria:

* Desire to take FZT 233 Effective Communication with Creative Drama in Health course at his own request.

  * Not wanting to participate in the study
  * Having a diagnosed psychological disorder and/or receiving psychological treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
interpersonal communication questionnaire | Change from Baseline interpersonal communication questionnaire at 14 weeks
  It is stated that the first four items are related to communication anxiety and the last four items are related to communication trust. Each item has a 5-point Likert scale between 1 = strongly disagree 5 = strongly agree. High values indicate poor communication
Jefferson Doctor Empathy Scale | Change from Baseline Jefferson Doctor Empathy Scale at 14 weeks
  The score range is 20-140, with higher average scores representing higher levels of empathy.

SECONDARY OUTCOMES:
Visual analog scale-communication | Change from Baseline Visual analog scale at 14 weeks
  A visual analog scale between 0 and 10 will be used to evaluate the communication that may occur when students go into clinical practice at the beginning and end of the term and when they meet the patient. Zero will be set to none, 10 will be set to the maximum I can think of.
Visual analog scale-anxiety/stress | Change from Baseline Visual analog scale at 14 weeks
  A visual analog scale between 0 and 10 will be used to evaluate the anxiety/stress that may occur when students go into clinical practice at the beginning and end of the term and when they meet the patient. Zero will be set to none, 10 will be set to the maximum I can think of.
Visual analog scale-motivation | Change from Baseline Visual analog scale at 14 weeks
  A visual analog scale between 0 and 10 will be used to evaluate the motivation that may occur when students go into clinical practice at the beginning and end of the term and when they meet the patient. Zero will be set to none, 10 will be set to the maximum I can think of.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided